CLINICAL TRIAL: NCT04767035
Title: A Pivotal Phase 1, Randomized, Single-Dose, 4-Period, Crossover Relative Bioavailability Study of MELT-100, IV Midazolam, and IV Ketamine Under Fasted Conditions in Healthy Volunteers
Brief Title: Relative Bioavailability Study of MELT-100, IV Midazolam, and IV Ketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melt Pharmaceuticals (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MELT-100-002
Record Dates: First submitted 2020-11-30; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Procedural Sedation
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: 4-period 4-arm crossover relative bioavailability
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MELT-100 3/25 (Active Comparator): MELT-100 3mg midazolam / 25 mg ketamine
  Interventions: Drug: midazolam / ketamine sublingual tablet
- MELT-100 2 x 3/25 (Active Comparator): MELT-100 2 doses of 3mg midazolam / 25mg ketamine
  Interventions: Drug: midazolam / ketamine sublingual tablet
- ketamine IV 18mg (Active Comparator)
  Interventions: Drug: midazolam / ketamine sublingual tablet
- Midazolam IV 3.5mg (Active Comparator)
  Interventions: Drug: midazolam / ketamine sublingual tablet

INTERVENTIONS:
Drug: midazolam / ketamine sublingual tablet — sublingual tablet

SUMMARY:
A Pivotal Phase 1, Randomized, Single-Dose, 4-Period, Crossover Relative Bioavailability Study of MELT-100, IV Midazolam, and IV Ketamine under Fasted Conditions in Healthy Volunteers

DETAILED DESCRIPTION:
A Pivotal Phase 1, Randomized, Single-Dose, 4-Period, Crossover Relative Bioavailability Study of 2 doses of 3.5mgMELT-100, IV Midazolam, and IV Ketamine 18mg under Fasted Conditions in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to understand and voluntarily consent to participation in this study and provides written informed consent before the start of any study-specific procedures.

  2. Healthy adult male or female at least 55 years of age. 3. Negative test for SARS-CoV2 (COVID-19) 4. Normally active and otherwise judged to be in good health on the basis of medical history and physical examination.

  5. Has vital signs (measured sitting after a minimum 3 minutes of rest) at Screening within the following ranges: heart rate: 40 to 100 bpm; systolic blood pressure (BP): 90 to145 mmHg; diastolic BP: 50 to 95 mmHg. Out-of-range vital signs may be repeated once.

  6. Has a body temperature ≤37.7 degrees C 7. Body weight at least 55 kg 8. Body mass index (BMI) 18.0 to 32.0 kg/m2 (inclusive) 9. Female subjects are eligible only if the following applies: Surgically sterile (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy), or postmenopausal (confirmed with serum FSH at Screening) 10. Male subjects must either be surgically sterile (vasectomy at least 3 months prior to first dose) or agree to use an acceptable method of birth control (see Section 4.4) from Screening through EOS.

  11. Is willing and able to remain in the study unit for the entire duration of each confinement period.

Exclusion Criteria:

* 1. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, ophthalmologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.

  2. Has a history of glaucoma, asthma, chronic obstructive pulmonary disease, or thyroid disease.

  3. History and/or family history of congenital long QT syndrome, unexplained syncope, or other additional risks for Torsade de Pointes, or sudden premature death.

  4. Clinically significant illnesses within 4 weeks of the administration of study medication (including flu, flu-like symptoms, diarrhea, vomiting, fever, sore throat) or acute illness at the time of either the pre-study medical evaluation or dosing.

  5. Has been in contact with someone within the last month who has tested positive for SARS-CoV-2.

  6. History of COVID-19. 7. Clinically significant surgery within 4 weeks prior to the administration of the study medication.

  8. Has participated in another clinical trial (randomized subjects only) within 30 days before the first dose of study medication.

  9. An active malignancy of any type or has been diagnosed with cancer within 5 years prior to Screening (excluding squamous or basal cell carcinoma of the skin).

  10. History or presence of allergic or adverse response to midazolam, ketamine, 11. Use of any over-the-counter (OTC) medication (including nutritional or dietary supplements, herbal preparations, or vitamins) within 14 days before the first dose of study medication until the EOS without evaluation and approval by the Investigator.

  12. Use of any prescription medication, except statin drugs or hormonal replacement therapy, from 14 days before the first dose of study medication until the EOS without evaluation and approval by the Investigator.

  13. Have had a depot injection or an implant of any drugs 3 months prior to administration of study medication.

  14. Has been treated with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) enzymes (e.g., barbiturates, phenothiazines, cimetidine, carbamazepine) within 30 days before the first dose of study medication, and that, in the Investigators judgment, may impact subject safety or the validity of the study results.

Specifically, the use of any drugs known to inhibit CYP2C9 and CYP3A4 enzymes (for example, amiodarone, fluconazole, ketoconazole, itraconazole, clarithromycin, ritonavir, erythromycin) or any drugs that are highly protein-bound (for example, warfarin, cyclosporine, amphotericin B) within 30 days prior to the first dose of study medication, and that in the Investigator's judgment may impact subject safety or the validity of the study results.

15. Blood or plasma donation within 30 days before the first dose of study medication until the EOS. It is recommended that blood/plasma donations not be made for at least 30 days after the EOS.

16. Has any prior history of substance abuse or treatment (including alcohol).

1. History of significant alcohol abuse within 6 months of Screening or any indication of the regular use of more than 2 units of alcohol per day

   (1 unit = 50 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
2. History of use of marijuana within 3 months of Screening or drugs such as cocaine, phencyclidine (PCP), within 1 year of Screening.

   17. Smoking or use of tobacco- or nicotine-containing products within 60 days before the first dose of study medication until the EOS Note: Nonsmokers are preferred for this study. 18. Any food allergy, intolerance, restriction, or special diet that, in the opinion of the Investigator, contraindicates the subjects participation in this study.

   19. Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.

   20. Consumption of beverages or foods that contain alcohol, poppy seeds, broccoli, Brussels sprouts, pomegranate, star fruit, char-grilled meat, or caffeine/xanthine from 48 hours before the first dose of study medication until the EOS.

   Subject must not consume grapefruit, orange, or apple juice from 7 days before the first dose of study medication until the EOS.

   Subjects will be instructed not to consume any of the above products; however, allowance for an isolated single incidental consumption may be evaluated and approved by the study Investigator based on the potential for interaction with the study drug.

   21. Engagement in strenuous exercise from 48 hours before the first dose of study medication until the EOS.

   22. A clinically significant abnormal finding on the physical examination, medical history, or clinical laboratory results at Screening.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Cmax | 24 hours
  Maximum Concentration
AUClast | 24 hours
  Area under the curve

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No